CLINICAL TRIAL: NCT00898274
Title: Antioxidant Enzymes and Oxidative DNA Damage in Subjects With 'High-Risk' for Prostate Cancer
Brief Title: Study of Blood Samples From Older Patients at High Risk of Developing Prostate Cancer and From Healthy Male Participants
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE11807; P30CA043703 (NIH); CASE11807 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Precancerous Condition; Prostate Cancer
Keywords: prostate cancer; high grade prostatic intraepithelial neoplasia
MeSH Terms: conditions — Precancerous Conditions; Prostatic Neoplasms | interventions — Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from patients at high risk of developing prostate cancer and from healthy male participants.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High risk for developing prostate cancer: Male subjects age 45-65 at high risk for developing prostate cancer.
  Interventions: Other: immunoenzyme technique; Other: laboratory biomarker analysis
- Healthy participants: Aged matched healthy participants
  Interventions: Other: immunoenzyme technique; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: immunoenzyme technique — Participants undergo blood sample collection. Samples are used to measure levels of antioxidant enzymes (i.e., glutathione, glutathione peroxidase, glutathione reductase, superoxide dismutase, and reduced glutathione) and biomarkers of oxidative stress and DNA damage in leukocytes (i.e., thiobarbituric acid reactive substances [TBARS] and 8-hydroxydeoxyguanosine). Samples are analyzed via antioxidant enzyme assay, TBARS assay, and enzyme-linked immunosorbent assay.
Other: laboratory biomarker analysis — Participants undergo blood sample collection. Samples are used to measure levels of antioxidant enzymes (i.e., glutathione, glutathione peroxidase, glutathione reductase, superoxide dismutase, and reduced glutathione) and biomarkers of oxidative stress and DNA damage in leukocytes (i.e., thiobarbituric acid reactive substances [TBARS] and 8-hydroxydeoxyguanosine). Samples are analyzed via antioxidant enzyme assay, TBARS assay, and enzyme-linked immunosorbent assay.

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients who are at high risk of developing prostate cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood samples from patients at high risk of developing prostate cancer and from healthy male participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether there are any changes in pro-oxidant-antioxidant profiles in patients who are at high risk for developing prostate cancer.
* To compare the profiles of these patients with those of healthy controls.

OUTLINE: Participants undergo blood sample collection. Samples are used to measure levels of antioxidant enzymes (i.e., glutathione, glutathione peroxidase, glutathione reductase, superoxide dismutase, and reduced glutathione) and biomarkers of oxidative stress and DNA damage in leukocytes (i.e., thiobarbituric acid reactive substances [TBARS] and 8-hydroxydeoxyguanosine). Samples are analyzed via antioxidant enzyme assay, TBARS assay, and enzyme-linked immunosorbent assay.

PROJECTED ACCRUAL: A total of 40 participants (20 at high risk for developing prostate cancer and 20 healthy controls) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patient at high risk for developing prostate cancer, due to 1 of the following risk factors:

    * Histologically confirmed proliferative inflammatory atrophy and/or high-grade prostatic intraepithelial neoplasia lesions accompanied by chronic intraprostatic inflammation
    * Abnormality observed during digital rectal exam or transrectal ultrasonography
    * Continued elevated age-adjusted prostate-specific antigen (PSA) meeting at least 1 of the following criteria:

      * Screening PSA > 4.0 ng/mL
      * Free PSA < 18%
      * PSA velocity > 0.75 ng/mL within the past year
  * Healthy volunteer meeting the following criteria:

    * Age-matched
    * Normal PSA level (≤ 2.1 ng/mL)
    * Normal digital rectal exam
    * No prostatitis or benign prostate hyperplasia
    * No urinary symptoms (diagnosed or undiagnosed)
* No diagnosis of cancer

PATIENT CHARACTERISTICS:

Patients and healthy controls:

* No chronic inflammatory conditions, especially those for which regular use of non-steroidal anti-inflammatory medications (NSAIDs) is prescribed/recommended, including any of the following:

  * Coronary heart disease
  * Chronic obstructive pulmonary disease (COPD)
  * Psoriasis
  * Pelvic inflammatory disease
  * Multiple sclerosis
  * Arthritis
  * Lupus
  * Hashimoto thyroiditis
  * Inflammatory bowel disease (i.e., ulcerative colitis or Crohn disease)

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or surgery to the prostate (healthy controls)

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Plasma levels of antioxidant enzymes as assessed by antioxidant enzyme assay, TBARS assay, and enzyme-linked immunosorbent assay | at time of study entry
  Blood (5ml) will be drawn from subjects for use in the various assays.
Oxidative DNA damage as assessed by antioxidant enzyme assay, TBARS assay, and enzyme-linked immunosorbent assay | at time of study entry
  Blood (5ml) will be drawn from subjects for use in the various assays.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Gupta, PhD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio